CLINICAL TRIAL: NCT06022588
Title: Heavy Isotope-labeled-butyrate and Glucose in Breath Testing to Detect Mesenteric Ischemia, a Proof-of-concept Study in Healthy Volunteers.
Brief Title: Chronic Mesenteric Ischemia Breath Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marco J. Bruno, Gastroenterologist, Erasmus Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL72878.078.20
Record Dates: First submitted 2023-07-26; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Chronic Mesenteric Ischemia
Keywords: Chronic mesenteric ischemia; Diagnostic; Breath test
MeSH Terms: conditions — Disease | interventions — Butyric Acid; Breath Tests; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 13C -butyrate control group (Placebo Comparator): 5 healthy volunteers performed the breath test without any psychical exercise
  Interventions: Drug: Sodium butyrate, 1-13C, 99%, Cambridge Isotope Laboratories, Inc.USA; Diagnostic Test: Breath test
- 13C -butyrate intervention group (Experimental): 5 healthy volunteers performed the breath test with psychical exercise - bicycle test
  Interventions: Drug: Sodium butyrate, 1-13C, 99%, Cambridge Isotope Laboratories, Inc.USA; Diagnostic Test: Exercise + breath test
- 13C -glucose control group (Placebo Comparator): 5 healthy volunteers performed the breath test without any psychical exercise
  Interventions: Drug: U-13C6, 99%; Cambridge Isotope Laboratories, Inc.USA; Diagnostic Test: Exercise + breath test
- 13C -glucose intervention group (Experimental): 5 healthy volunteers performed the breath test with psychical exercise - bicycle test
  Interventions: Drug: U-13C6, 99%; Cambridge Isotope Laboratories, Inc.USA; Diagnostic Test: Exercise + breath test

INTERVENTIONS:
Drug: Sodium butyrate, 1-13C, 99%, Cambridge Isotope Laboratories, Inc.USA — a solution containing butyrate of which 12C of the last 4 carbon positions of butyrate were replaced by 13C butyrate. Participants received 0.80 gram 13C-butyrate (7.3 mMol butyrate / 29 mMol 13C) dissolved in 50 mL water at baseline
  Other Names: 13C butyrate
  Arms: 13C -butyrate control group; 13C -butyrate intervention group
Drug: U-13C6, 99%; Cambridge Isotope Laboratories, Inc.USA — a glucose solution in which all six 12C carbons were replaced by 13C D-Glucose. Participants received 0.75 gram 13C-glucose (4.2 mMol D-glucose/ 25 mMol 13C) dissolved in 50 mL water at baseline
  Other Names: 13C glucose
  Arms: 13C -glucose control group; 13C -glucose intervention group
Diagnostic Test: Breath test — Breath tests were performed at the following time points baseline, 0.5, 1, 1.25 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5 and 4 hours after ingestion of 13C-butyrate and 13C-glucose. Breath samples were obtained by blowing a single breath of air through a straw into a test tube. Two breath samples were collected at all mentioned time points. Measurement of 13CO2 is performed using mass spectrometry (IDMicro Breath, Compact Science Systems, Newcastle-Under-Lyme, United Kingdom) using procedures described earlier for galactose and methacetin breath tests, and expressed as an absolute increase in the 13CO2-to-12CO2 ratio in delta permil (δ‰).
  Arms: 13C -butyrate control group
Diagnostic Test: Exercise + breath test — The intervention groups performed a standardized bicycle ergometer exercise test of 30 minutes and semi-continuous peripheral blood lactate monitoring. The bicycle ergometer protocol consists of three phases. The first 10 minutes of exercise was used to gradually increase the workload until submaximal exercise intensity was reached which is defined as a circulating blood lactate level between 3 and 5.5 mmol/L. From minute 10 to 20 submaximal exercise intensity was maintained by adjusting the workload based on lactate measurements. Minute 20 to 30 was used to reach maximal exercise intensity, the workload was increased by 10% of the submaximal workload until exhaustion
  Arms: 13C -butyrate intervention group; 13C -glucose control group; 13C -glucose intervention group

SUMMARY:
Background and aims:

A gold standard diagnostic test to diagnose chronic mesenteric ischemia is currently lacking. Isotope labelled-butyrate and glucose breath testing could theoretically quantify mucosal oxygen consumption and thereby detect ischemia, since oxygen is needed to absorb and metabolize butyrate and glucose, and distinguish aerobic/anaerobic intestinal epithelial metabolism. Here we aim to test this notion and compare results to conventional biomarkers.

Methods:

Healthy volunteers were randomized into two control groups and two intervention groups, each consisting of five volunteers receiving either oral 13C -butyrate or 13C -glucose. The control groups performed breath tests without any physical exercise. The intervention groups performed a 30 minutes standardized bicycle exercise test, which has been proven to elicit mesenteric ischemia. Breath samples of expired 13CO2 were collected during a period of 4 hours and results were contrasted to measurements of biomarkers in peripheral blood.

DETAILED DESCRIPTION:
Even as chronic mesenteric ischemia (CMI) is the most common vascular disorder involving the mesenteric arteries, accounting for 2% of all revascularization procedures, it remains an underdiagnosed condition. CMI is an invalidating disease that causes severe complaints of post-prandial abdominal pain, food fear and weight loss. Diagnosis of CMI remains difficult since no gold standard diagnostic test exists, the presumptive diagnosis of CMI is currently confirmed when a patient experiences relief of symptoms after revascularization. For making treatment decisions, clinicians rely on a consensus diagnosis, based on clinical history, presence of mesenteric artery stenosis on abdominal imaging, and, in dedicated centers, the outcome of a functional test, such as visible light spectroscopy (VLS) or tonometry. The diagnostic accuracy of this consensus diagnosis is unstatisfactory, since clinical improvement is achieved in only 73% of patients with a consensus diagnosis of CMI based on a single mesenteric artery stenosis. Per extenso in the remaining 27% treatment was initiated in patients not suffering from CMI. Stressing the need for a reliable diagnostic test to identify patients with CMI.

In the intestinal epithelium the most important substrate for mitochondrion-dependent ATP production, and by consequence as the source for CO2 release is butyrate, a small chain fatty acid produced by the intestinal microflora. Under ischemic conditions, butyrate can no longer be metabolized. The most straight forward biochemical pathway to cope with this situation is a switch in cellular metabolism to anaerobic glycolysis. In this process glucose is metabolized to pyruvate, producing two ATP molecules, providing an oxygen independent pathway for maintaining ATP production, but also resulting in the reduction of NAD+ molecules into NADH+. To maintain ATP production, pyruvate will undergo a process called fermentation resulting in the production of lactate in which NADH+ is recycled back to NAD+ so that glycolysis can continue. Upon subsequent transport via the blood, lactate is cleared in the liver and the resulting CO2 will leave the body via the lungs. Hence theoretically measuring the shift from butyrate towards glucose metabolism, which occurs in enterocytes under anaerobic conditions, could be a method to detect mucosal ischemia.

This multi-center randomized interventional proof of principal study explored the possibility to quantify mucosal oxygen content by labeled-butyrate and labelled-glucose breath testing as a potential test to diagnose CMI. Since both substrates are dependent on oxygen to be metabolized, it is expected that subjects with low mucosal oxygen concentrations will metabolize less butyrate and glucose compared to subjects with normal mucosal oxygen concentrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers without any gastrointestinal complaints

Exclusion Criteria:

* pregnant woman

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The median concentrations of measured 13CO2 | At the following time points; baseline, 0.5, 1, 1.25 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5 and 4 hours (total of 12 time points) after ingestion of 13C-butyrate or 13C-glucose.
  The median concentrations of measured 13CO2 at each time point where compared within the four groups and statistically tested with a Mann - Whitney U test.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, prof., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center - Department of Gastroenterology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT06022588/Prot_SAP_000.pdf